CLINICAL TRIAL: NCT04072185
Title: CHANGES IN THE EMOTIONAL STATE, QUALITY OF LIFE AND SOCIAL SUPPORT AFTER A PROGRAM OF PHYSICAL ACTIVITY IN THE ELDERLY PEOPLE: RANDOMIZED MULTI-CENTER CLINICAL TRIAL
Brief Title: PHYSICAL ACTIVITY AS A MEASURE OF IMPROVING THE EMOTIONAL STATE AND SOCIALIZATION IN THE ELDERLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI 19/031-P
Record Dates: First submitted 2019-07-19; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Depression; Anxiety; Social Isolation
Keywords: Physical activity; Primary Care; elderly people; anxiety; depression; social isolation
MeSH Terms: conditions — Depression; Anxiety Disorders; Social Isolation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized, two-group clinical trial, of 1 year follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity group (Experimental)
  Interventions: Other: Physical activity
- Control group (No Intervention)

INTERVENTIONS:
Other: Physical activity — TThe intervention group will participate in a group physical activity program for 4 months. It will consist of 60 minutes of walking sessions 2 days a week. The sessions will be directed by two referents of each primary care center. Also once a month, coinciding with the walk, you will visit some sociocultural municipal equipment to promote a community connection.
  Arms: Physical activity group

SUMMARY:
Background: Social isolation, loneliness and anxiety-depressive states are emerging health conditions in the elderly of our society. This situation is related to higher morbidity and mortality. There is a growing need to determine effective interventions that address these situations, since sometimes pharmacological options are limited in these patients. Physical activity (AF) and social relationships in the elderly are linked to physical and mental health. Being able to do some physical or recreational activity will help them face this stage of life with more optimism and relate to others in a healthy and independent way, however, few studies have evaluated their effectiveness in our territory.

* Objectives: To evaluate whether a 4 month AF group program and the visit to know socio-cultural entities improve the emotional, social and quality of life situation in a sample of people over 64 years of age with anxiety, depression, social isolation or solitude And measure whether adherence to AF and the linkage to sociocultural entities is maintained after the intervention has taken place.
* Methodology:

Design: Multicentre, randomized, two-group clinical trial, of 1 year follow-up. Study population: Patients over 64 years of age assigned to primary care teams (EAP) from different locations: Sant Joan de Vilatorrada, Súria and Manresa 2.

Inclusion criteria: To meet criteria of depression or anxiety at the time of the study, score> 12 on the Beck Depression Scale and / or score> 10 on the GAD-7 Scale (General Anxiety Disorder) and that Present a score <32 on the steps of DUKE-UNC-11.

A randomization of between 44 and 56 patients will be performed at each participant EAP. Half will be allocated to the control group (GC) and half to the intervention group (GI).

The intervention group will participate in a group AF program for 4 months. It will consist of 60 minutes of walking sessions 2 days a week. Also once a month, coinciding with the walk, you will visit some sociocultural municipal equipment to promote a community connection.

. Main measures: Response to the intervention or clinical remission of depression (Escalera de Beck), and / or anxiety (Escala GAD-7), improvement of social support (DUKE-UNC) and quality of life (EuroQol) . Secondary measures: Adherence to the AF (VREM questionnaire (Spanish Reduced Version of the Minnesota Free Time Questionnaire in Minnesota)), and linkage to sociocultural entities once the intervention has been completed. The assessments will be made at 0, 4, 8 and 12 months.

DETAILED DESCRIPTION:
BACKGROUND AND CURRENT STATUS OF THE SUBJECT:

In our society, thanks to medicine and development, the proportion of the elderly population tends to increase every year. The percentage of people over 64 years of age in 2017 in Spain was 18.8%, and is expected to continue to increase to 34.6% in 2066, according to the National Statistics Institute projection (1).

Social isolation, loneliness and anxiety-depressive states are emerging health conditions in the elderly in our society. As much in adult population as in old population noninstitutionalized it has been verified that to have little social support is related to a worse mental health. According to the European Health Survey in Spain carried out by the Ministry of Health, Consumption and Social Welfare of 2017, the prevalence of depression and chronic anxiety were in subjects of 65-74 years of 10.64% and 8.25% , from 75 to 84 years of 13.73% and 9.49% and over 85 years of 11.36% and 6.68% (2). This situation is related to higher morbidity and mortality. There is a growing need to determine effective interventions that address these conditions, since sometimes pharmacological options are limited in these patients.

For decades it has been known that social relationships are linked to physical and mental health. A satisfying social network promotes healthy behaviors and habits. Social support especially protects the elderly from loneliness (3) and from depression (4). In particular, it can have a beneficial impact on mental health problems and psychological distress among older adults (5).

Also AF in the elderly has multiple advantages, not only at the physical level but also at the emotional level (6-8), several studies show that physical or leisure activities reduce loneliness (9), depression (10- 14), anxiety (15) and are associated with better mental health (16, 17). According to Guszkowska (18), the AF's benefits of anxiety, depression and irritability are especially high in those who start from high levels of anxiety and depression. The type of AF that causes major improvements is those based on cyclical aerobic activities (walking, swimming or cycling) from moderate to low intensity. This statement is aligned with the position of the American College of Sports Medicine, which recommends AF for the larger populations and affirms that regular AF can minimize the physiological and psychological effects of a sedentary lifestyle time that increases the expectations of life (19) and the quality of life (20). Being able to do some physical or recreational activity will help them face this stage of life with more optimism and relate to others in a healthy and independent way (21), however, few studies in our territory have evaluated their effectiveness.

HYPOTHESIS

* The AF improves the emotional, social and quality of life situation in subjects over 64 years of age with problems of anxiety, depression, social isolation or loneliness.
* The intervention group remains more active than the control group.
* The intervention favors maintaining the AF for a long period.
* The intervention group is more linked to sociocultural entities than the control group.

TARGETS

Main objective:

-To evaluate if the AF improves the emotional, social and quality of life situation in a sample of people over 64 years of age with problems of anxiety, depression and little social social support.

Secondary goals:

* Evaluate whether the intervention of an AF program for 4 months keeps improving the emotional, social and quality of life situation in a sample of people over 64 years of age with anxiety, depression, social isolation or loneliness at 8 and 12 months of the intervention.
* Measure if the adherence to the AF is maintained after the intervention has taken place at 8 and 12 months.
* Measure if the link to sociocultural entities is created and maintained once the intervention has been carried out at 4, 8 and 12 months
* Evaluate the satisfaction of the users after the intervention at 4 months.

METHODOLOGY Design: Multicentre, randomized, two-group clinical trial, of 1 year follow-up. Study population: Patients over 64 years of age assigned to primary care teams (EAP) from different locations: Sant Joan de Vilatorrada (12,721 assigned), Súria (8,956 assigned), Manresa 2 (23,351 assigned). With this representativeness of territories, patients living in urban, semi-urban and rural areas will be able to study. Subsequently, the participation of other SAP teams will be attempted.

Inclusion criteria: Meet the criteria of depression or anxiety at the time of the study, score> 12 on the Beck Depression Scale (BDI-II) and / or score> 10 on the GAD-7 Scale (General Anxiety Disorder) and that they score <32 on the back of DUKE-UNC-11. Possibility to follow a year by the same primary care team. At least read and write Spanish or Catalan.

Exclusion criteria. Diagnosis of dementia or moderate cognitive impairment. Greater depression (BECK scale score> 28). Dependency disorders due to abuse of alcohol or other drugs. You are receiving some psychological therapy from the Center for Reference Mental Health. Physical illness at an advanced stage. Present any physical, mental or temporary limitations to be able to walk 1 hour a day two days a week. That they have not signed the informed consent.

Show and recruitment: Each participating Primary Care Team (EAP) will be randomized between 44 and 56 patients. Half will be allocated to the control group (GC) and half to the intervention group (GI). The recruitment will be consecutive in each EAP.

The professionals participating in the study will consult the database of the Computerized Clinical History of Catalonia (ECAP) through the consultation form of their quotas (Dbsform), in order to obtain the lists of patients that meet the inclusion criteria (have the active diagnosis of depression or anxiety and have little social support). Subsequently, your doctor or nurse will make the selection of the patients and will contact them to offer them the possibility to participate in the study and, in case they accept, they will be grouped in their CAP to explain In detail, study and sign informed consent, an interview will be followed and the questionnaires will be administered to assess whether they meet the inclusion criteria. They will finally be assigned to Control group or intervention randomly and anonymously using a statistical program.

Sample size: The sample size for independent groups was estimated, capable of detecting differences of two points in the average score of the Depression of Beck and GAD-7 and 7 points in the scale of social support of DUKE-UNC-11. A control has been assigned for each case, assuming a statistical power of 80% with a confidence interval of 95%. Between 146 and 162 patients would be needed and for reasons of convenience three groups of 50 patients each will form in each EAP, 25 of which will be in the intervention groups and 25 in the control units.

Variables and measurement methods:

Variables main results:

1. Clinical remission of depression and / or response to the intervention once the intervention has been completed, at 4 months after the start of the study. Clinical remission is considered: Beck scale score (BDI-II) <12 points (Riedel 2010) and response to the intervention: reduction of the basal score. The Beck Depression Inventory is an auto-applied questionnaire of 21 items with four response alternatives, sorted according to the severity of the symptoms it refers to (range 0 to 3; range score from 0 to 63 scale). The version adapted to Spanish by Sanz (2003) will be used.
2. Remission of the anxiety clinic and / or response to the intervention once the intervention has been completed, at 4 months after the start of the study. Clinical remission is considered: scaling of the GAD-7 scale (General Anxiety Disorder) <10 points and response to the intervention: reduction of the score compared to basal. The GAD-7 scale is simple and self-administrable, it has 7 items of anxiety symptoms on a Likert scale on the presence of the symptom in the last two weeks ("nothing at all", "several days", "more than half of the days "and" almost every day ") that score from 0 to 3, where the maximum score is 21. A score greater than or equal to 10 is indicative of anxiety disorders, achieving a sensitivity of 89% and a specificity of 82 %. This scale has been validated in Spanish by García-Campayo (2010).
3. Improvement of social support once the intervention has finished 4 months after the start of the study. Social support improvement is considered a decrease in the score in the DUKE-UNC-11 social support questionnaire with respect to the basal, and good social support with a score <32 points. This instrument was designed to measure functional social support perceived by Broadhead and validated for the Spanish population by Bellón et al. (1996). This is a self-administered 11 item instrument, uses a Likert type response scale with scores from 1 to 5, stands out for its simplicity and brevity, evaluates the perceived social support, evaluates the confidential social support (possibility of have people to communicate) and affective social support (demonstrations of love, affection and empathy). In the Spanish version, a cut-off point was chosen in the 15th percentile, which corresponds to a score <32, to divide the subjects into two groups (normal or low support).
4. Improved quality of life once the intervention has been completed at 4 months after the start of the study. Quality of life improvement is considered a decrease in the score in the EuroQol questionnaire (EQ-5D) with respect to basal.

Secondary result variables:

1. Clinical remission of depression and / or response to the intervention at 8 and 12 months.
2. Clinical remission of anxiety and / or response to the intervention at 8 and 12 months.
3. Improvement of the situation / social perception (DUKE-UNC Social Welfare Questionnaire) at 8 and 12 months.
4. Improved quality of life measured through EuroQol (EQ-5D) at 8 and 12 months.
5. Result variables that measure feasibility in the intervention group:

   * Satisfaction with the intervention: A patient satisfaction survey will be carried out at the end of the intervention, with 5 items and Likert scale of 4 categories.
   * Adherence to the intervention: for each GI patient the number of sessions attended will be collected. A variable of adherence to the intervention will be calculated: attend 75% or more of the sessions, attend less.
   * Adherence to AF post intervention through the VREM Questionnaire (Reduced Spanish version of the AF time questionnaire in Minnesota)). The assessments will be made at 0, 4, 8 and 12 months.
6. Linking to sociocultural entities once the intervention has been completed. The assessments will be made at 0, 4, 8 and 12 months.

Variables that can act as confusers or modifiers of the effect:

1. Pharmacological treatment. The DDD (defined daily dose) must be calculated for each active ingredient in the follow-up period, taking into account the number of days, the dose provided and the route of administration of the drug. The active principles that will be registered will be those belonging to the following groups: antidepressants, anxiolytics.
2. Participation in other mental health therapies, taught by a psychologist, psychiatrist. Patients included in the therapies of the reference mental health centers will be excluded.
3. Prior participation in some AF activity on a regular basis: yes / no. Socio-demographic variables: Sex, age, marital status, live life (yes / no), educational level (without studies / incomplete primary / full primary / high school / higher education). Reference primary care team: rural (assigned to a doctor's office) / semi-urban (assigned to an AP center in a population <15,000 inhabitants) / urban (assigned to an AP center with a population of 15,000 or more).

Intervention:

The intervention group will participate in a group AF program for 4 months. It will consist of 60 minutes of walking sessions 2 days a week. The sessions will be directed by two referents of each CAP, which will carry an application to the mobile (type STRAVA), to control the distances recurred from each session. Also once a month, coinciding with the walk, you will visit some sociocultural municipal equipment to promote a community connection.

Data collection:

In the field work, different groups of professionals participate:

* Professional recruiters: doctor and / or nurse to which the patient is assigned.
* Researcher in charge of the random allocation of patients: not linked to any EAP. Perform the random assignment once all the patients required in each team have consented to participate.
* Evaluators: carry out baseline interviews at 4, 8 and 12 months, without knowing which group the patient belongs to.
* Professionals that will accompany the walks: two for each EAP.
* Professionals from sociocultural centers.

The external evaluator will be in charge of collecting the results of the self-administered scales previously mentioned in paper. These stairs will be in a unique place that only this reviewer will have access to. They will be read with automatic reading with the identifier of the survey using the Teleform Elite v 8.2 reading software.

DATA ANALYSIS:

Initially, the sociodemographic characteristics of the two groups will be described. For the description of qualitative variables, percentages and for quantitative, standard averages and averages, ranges and 25-75 percentiles will be used.

Previous to the intervention, baseline scores on the selected scales after randomization of the patients will be compared to verify that there are no significant differences. After the intervention, the average scores of the different scales in both groups will be compared independently, and for the different periods of post-intervention time, using the Student test for matched samples in case of normality adjustment or the Mann-Whitney U if the distribution was not normal. A secondary analysis, through multiple regression, will be carried out, including sociodemographic and confusing variables, for the variable of clinical remission of depression Yes / No (Yes: Beck scale <12), for the clinical remission variable of anxiety Yes / No (Yes: GAD-7 <10) and for the social support variable Yes / no (Yes: DUKE-UNC-11> 32).

The results showing differences with a p <0.05 will be considered significant. For statistical analysis, it was used in program SPSS v. 18.

ETHICAL CONSIDERATIONS:

In accordance with Law 14/2007 of July 3, of biomedical and human rights research (BOE of July 4, 2007), all recruited patients will be informed verbally and in writing of the objectives, methodology, tests and interventions that can be received if they participate in the study. It will be included to those who sign informed consent in writing. The document will be written in a language that the patient can understand. The protocol has been approved by the Ethical Committee of Clinical Investigation of the JGol Idiap. The researchers undertake to maintain the confidentiality of the data. If the effectiveness of the intervention is shown, the control group will receive the same group intervention once the study has finished.

ELIGIBILITY:
Inclusion Criteria:

* score > 12 on the Beck Depression Scale (BDI-II)
* and / or score > 10 on the GAD-7 Scale (General Anxiety Disorder)
* and / or score < 32 on the back of DUKE-UNC-11.

Exclusion Criteria:

* Diagnosis of dementia or moderate cognitive impairment.
* Greater depression (BECK scale score> 28).
* Dependency disorders due to abuse of alcohol or other drugs.
* Participate in a therapy group of the hospital's psychiatry department.
* Physical illness at an advanced stage.
* Present any physical, mental or temporary limitations to be able to walk 1 hour a day two days a week.
* Not having signed the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-03-14 (Estimated); Study Completion 2020-09-14 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline The Beck Depression Inventory score | 4, 8 and 12 months after starting the study.
  Clinical remission is considered: Beck scale score (BDI-II) <12 points (Riedel 2010) and response to the intervention: reduction of the basal score.
Change from Baseline General Anxiety Disorder-7 scale score | 4, 8 and 12 months after starting the study.
  Clinical remission is considered: scaling of the GAD-7 scale (General Anxiety Disorder) <10 points and response to the intervention: reduction of the score compared to basal
Change from Baseline DUKE-UNC-11 social support questionnaire score | 4, 8 and 12 months after starting the study.
  Social support improvement is considered a decrease in the score in the DUKE-UNC-11 social support questionnaire with respect to the basal, and good social support with a score <32 points.
Change from Baseline EuroQol quality of life questionnaire score | 4, 8 and 12 months after starting the study.
  Quality of life improvement is considered a decrease in the score in the EuroQol questionnaire with respect to basal.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Mendioroz, MD, Study Chair — Institut Català de la Salut
Locations (1):
- Sant Joan de Vilatorrada Primary Care Center, Sant Joan de Vilatorrada, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No